CLINICAL TRIAL: NCT02460432
Title: A Prospective, Randomized, Single Blind Study to Evaluate the Effectiveness and Safety Comparing Niti-S Mira-Cover III Biliary Stent With ComVi Biliary Covered Stent in Patients With Malignant Biliary Obstruction
Brief Title: Comparison of Drug Eluting Stent and Covered Metal Stent in Malignant Biliary Obstruction (MIRA III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRA-003
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Biliary Neoplasms; Biliary Obstruction; Pancreatic Neoplasms
Keywords: Drug-eluting Biliary stent; Covered metalic stent
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-eluting metal Stent (Experimental): Niti-S Mira-Cover III Biliary Stent (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Paclitaxel-eluting metal Stent
- Covered Metal Stent (Active Comparator): ComVi Biliary Covered Stent (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Covered Metal Stent

INTERVENTIONS:
Device: Paclitaxel-eluting metal Stent — Insertion of Niti-S Mira-Cover III Biliary Stent using ERCP
  Arms: Paclitaxel-eluting metal Stent
Device: Covered Metal Stent — Insertion of ComVi Biliary Covered Stent using ERCP
  Arms: Covered Metal Stent

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of Niti-S Mira-Cover III Biliary Stent with Comvi Biliary Covered Stent for the treatment of malignant biliary obstruction.

DETAILED DESCRIPTION:
In patients with malignant biliary obstruction, endoscopic placement of biliary stents offers similar technical success rates. Endoscopic retrograde cholangiography (ERCP)-guided stent placement has become the preferred approach to palliate malignant biliary obstruction. The major mechanisms of self-expandable metallic stent (SEMS) occlusion are tumor ingrowth, tumor overgrowth, and epithelial hyperplasia. These mechanisms provide the rationale for developing a drug-eluting stent in order to improve stent patency. Limited data exist regarding outcomes of paclitaxel-eluting stents in malignant biliary obstruction. This study is to prospectively compare the effectiveness and safety of paclitaxel-eluting covered metal stent and covered metal stent for the treatment of malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 19 years of age
* Malignant mid or distal biliary obstruction
* Unresectable cancer
* Estimated survival greater than or equal to 3 months (Karnofsky score ≥ 60)
* Patient willing to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

* Patients who had undergone surgical biliary drainage
* Severe bleeding disorder (e.g. coagulopathy)
* Polypoid lesion or intra-abdominal abscess
* Female of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12-26 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
Cumulative stent patency during 6months after stent placement | 6 month
  Stent patency is defined as absence of stent obstruction and confirmed by computed tomography (CT) or ERCP.

SECONDARY OUTCOMES:
Stent migration | 6 month
  Stent migration is defined as an obvious dislodgement from the intended and original implant position and confirmed by radiography, CT, or ERCP.
Secondary stent insertion due to recurrent biliary obstruction | 6 month
Mean survival | 6 month
Adverse events | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Lee, Ph.D MD, Study Chair — Gangnam Severance Hospital; Kyu Taek Lee, Ph.D MD, Principal Investigator — Samsung Medical Center; Sang Hyub Lee, Ph.D MD, Principal Investigator — Seoul National University Hospital; Don Haeng Lee, Ph.D MD, Principal Investigator — In Ha University Hospital; Jung Sik Choi, Ph.D MD, Principal Investigator — Inje University
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan, Bokji-ro Busanjin-gu
  - Seoul National University Hospital, Seoul, Haehak-ro Jongno-gu
  - In Ha University Hospital, Incheon, Inhang-ro Jung-gu
  - Samsung Medical Center, Seoul, Irwon-Dong, Gangnam-Gu
  - Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
February 12, 2016

REFERENCES:
- [Derived] Jang SI, Lee KT, Choi JS, Jeong S, Lee DH, Kim YT, Lee SH, Yu JS, Lee DK. Efficacy of a paclitaxel-eluting biliary metal stent with sodium caprate in malignant biliary obstruction: a prospective randomized comparative study. Endoscopy. 2019 Sep;51(9):843-851. doi: 10.1055/a-0754-5763. Epub 2018 Nov 9. PMID 30414164